CLINICAL TRIAL: NCT01089374
Title: A Prospective Study of Partial Breast Adjuvant Radiation Therapy After Resection of Borderline and Malignant Phyllodes Tumors
Brief Title: Phyllodes Tumor Partial Breast Radiation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low disease incidence rate
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., MD, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0929
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Phyllodes Tumor
Keywords: Phyllodes
MeSH Terms: conditions — Phyllodes Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Partial breast radiation after lumpectomy (Other): Radiation per NSABP B-39/R0413 protocol.
  Interventions: Radiation: Partial breast radiation after lumpectomy

INTERVENTIONS:
Radiation: Partial breast radiation after lumpectomy — Radiation therapy will be administered in the vicinity of the center where the surgical resection was performed. Adjuvant radiation must start within 12 weeks of breast excision or re-excision. The radiation oncologist can choose between two methods of partial breast irradiation (PBI): external beam partial breast radiation or Mammosite® brachytherapy, based on radiation oncologist and patient preference. Radiation will be administered per guidelines used in the NSABP B-39/RTOG 0413 protocol.

SUMMARY:
In 2008 a research study conducted by Dr. Barth involving 46 women determined that whole breast radiation therapy performed after a lumpectomy of borderline and malignant phyllodes tumors decreases rate of recurrence. None of the 46 participants developed a local recurrence.

Based on information we have learned from research studies, we recommend whole breast radiation therapy for women with malignant and borderline phyllodes tumors after they receive a lumpectomy.

New methods for delivering breast radiotherapy are being developed that allow radiation to be delivered solely to the site of the surgical resection. This is called partial breast radiation. The main advantage of partial breast radiation is that it simplifies treatment for the patient. Radiation is delivered twice a day for 5 days, rather than 5 days per week for 6 weeks. The main concern is that partial breast radiation might miss other sites of breast cancer in the breast receiving the radiation.

Evidence is accumulating from research studies that partial breast radiation therapy after surgical removal of the more common type of breast cancer, invasive ductal carcinoma, the breast results in rates of local recurrence that are comparable to those seen after whole breast radiation therapy.

In contrast to patients with invasive ductal cancers of the breast, it is very rare for patients to have phyllodes tumors that appear in more than one area of the breast. Review of research data determined that cancer recurrences seen in patients with phyllodes tumors that had undergone lumpectomies were almost always at the original tumor site. Therefore, partial breast radiation is likely to be as effective as whole breast radiation therapy after resection of malignant phyllodes tumors.

The purpose of the study is to determine what the chances are that a phyllodes tumor will recur in the breast when the breast is treated with partial breast radiation therapy after a lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of phyllodes tumor of borderline or malignant grade, as first defined by Pietruszka and modified by Azzopardi and adopted by the World Health Organization (1,2,17):

  * Borderline malignant: 5-9 mitoses/10 HPF, pushing or infiltrating margins, 2+ (moderate) stromal cellularity and atypia.
  * Malignant: 10 or more mitoses / 10 HPF, predominantly infiltrating margins, usually 3+ (severe) stromal cellularity and atypia but occasionally 2+.
* The tumor has been excised with a breast-conserving resection and there is no tumor seen at any of the margins of the resection.
* No prior breast carcinoma or ductal carcinoma in situ in the ipsilateral breast. Patients with a local recurrence of a previously excised phyllodes tumor are eligible if the recurrence is in the area of the previous excision.
* No history of irradiation of the ipsilateral breast.
* No evidence of other areas worrisome for cancer on physical examination and mammography of the ipsilateral breast.
* Age >18 years.
* Informed consent.
* Documentation that either:

  1. the patient's medical insurance company has certified that they will pay for the cost of radiation therapy treatments, or
  2. a letter from the patient indicating that they explicitly understand the costs of radiation therapy and that the sponsor (Principal Investigator) of this study will not be held responsible for these costs.

Exclusion Criteria:

* Histologically positive margins.
* Breast carcinoma or ductal carcinoma in situ in the ipsilateral breast.
* A history of irradiation to the ipsilateral breast.
* Pregnancy. A urine pregnancy test will be performed on each fertile premenopausal female prior to entry into the study. Patients with childbearing potential must employ effective contraception during the radiation therapy.
* A radiation planning CT scan which demonstrates a target lumpectomy cavity that is not clearly delineated or a target lumpectomy cavity/whole breast reference volume > 30%.
* Unacceptable radiation therapy quality assurance parameters, as defined in Section 5 of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01-12 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Barth, JR, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Historical controls were not enrolled as part of this study. Information regarding the historical controls can be found under NCT00003404.
Groups:
- Historical Control: Historical controls treated with whole breast radiation therapy after breast conserving resection with negative margins. Information regarding the historical controls can be found under NCT00003404.
Period: Overall Study
Arm/Group | Partial Breast Radiation After Lumpectomy | Historical Control
Started | 11 | 46
Completed | 1 | 46
Not Completed | 10 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study closed early - low accrual | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Historical Control: Historical controls treated with whole breast radiation therapy after breast conserving resection with negative margins
- Total: Total of all reporting groups
Arm/Group | Partial Breast Radiation After Lumpectomy | Historical Control | Total
Number analyzed (Participants) | 11 | 46 | 57
Age, Continuous [Mean (Full Range); unit: years] | 46 [19 to 64] | 49 [18 to 76] | 47.5 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 46 | 57
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 0 | 9
  Unknown or Not Reported | 1 | 46 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 0 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 46 | 47
Region of Enrollment [Number; unit: participants]
  United States | 11 | 46 | 57

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participants With Local Recurrence up to 10 Years
Description: The primary objective is to determine the local recurrence rate for patients with borderline or malignant phyllodes tumors treated with breast conserving resection with negative margins and adjuvant partial breast radiation therapy. Recurrence rate is measured by occurrence of biopsy proven recurrences during follow up, up to 10 years following patient enrollment.
Time Frame: up to 10 years
Population: The following participants did not complete 10 years of follow up and were followed until the time points listed below:
  1. participant lost to follow up after 6 months
  2. participants lost to follow up after 1 year
  1 participant withdrew after 9 years 6 participants remained on study until early study closure they were at the following time points at closure: 2 participants 4.5 years
  1 participant 5 years
  1 participant 6 years
  1 participant 8 years
  1 participant 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Radiation After Lumpectomy
Number analyzed (Participants) | 11
Participants | 0

2. Secondary Outcome: Rate of Participants With Local Recurrence After Radiation Compared to Historic Controls
Description: The secondary objective is to compare the local recurrence rate observed after partial breast radiation therapy with that observed in historical controls treated with whole breast radiation therapy after breast conserving resection with negative margins. This is measured by occurrence of biopsy proven recurrence up to 10 years after participant enrollment.
Time Frame: up to 10 years
Population: The following participants did not complete 10 years of follow up and were followed until the time points listed below:
  1. participant lost to follow up after 6 months
  2. participants lost to follow up after 1 year
  1 participant withdrew after 9 years 6 participants remained on study until early study closure they were at the following time points at closure 2 participants 4.5 years
  1 participant 5 years
  1 participant 6 years
  1 participant 8 years
  1 participant 9 years
Measure: Count of Participants; unit: Participants
Groups:
- Historical Controls: Historical controls treated with whole breast radiation therapy after breast conserving resection with negative margins.
Arm/Group | Partial Breast Radiation After Lumpectomy | Historical Controls
Number analyzed (Participants) | 11 | 46
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All patients will be encouraged to perform monthly breast self examination and will be followed with physical exams of the affected breast by their surgeon or radiation oncologist. These physical exams should occur every 6 months (+/- 3 months) after the initial resection through year 5 ( ie. at 6,12,18,24,30,36,42,48,54,and 60 months) and then every 12 months (+/- 3 months) years 5 through 10 (ie. 72, 84, 96,108 and 120 months).
Description: These physical exams should occur every 6 months (+/- 3 months) after the initial resection through year 5 ( ie. at 6,12,18,24,30,36,42,48,54,and 60 months) and then every 12 months (+/- 3 months) years 5 through 10 (ie. 72, 84, 96,108 and 120 months). Information relating to adverse events and serious adverse events for the historical controls can be found under NCT00003404.
Arm/Group | Partial Breast Radiation After Lumpectomy
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial Breast Radiation After Lumpectomy (N=11)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT01089374/Prot_SAP_000.pdf